CLINICAL TRIAL: NCT06684496
Title: Strength Training and Thoracic Aorta Dilatation: an Echocardiographic Cross-sectional Study
Brief Title: A Study of High-intensity Strength Training and Thoracic Aorta Dilatation
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Darrell B. Newman, Principal Investigator, Mayo Clinic
Other Study IDs: 24-007099
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Thoracic Aorta Dilatation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to describe the prevalence of thoracic aorta dilatation among a group of older (age > 35 years), experienced weightlifters (>5 years of weightlifting experience). The secondary aim of this study is to report the prevalence of thoracic aorta dilatation among 3 different groups of weightlifters (body builders, cross-fit athletes, and power lifters).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 35
* ≥5 years of weightlifting experience

Exclusion Criteria:

* Age < 35
* < 5 years of weightlifting experience
* personal history of thoracic aorta dilatation/aneurysm/dissection

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is power lifters (n=15), body builders (n=15), and cross-fit (n=15) athletes age 35 years or older with at least 5 years of consistent weight training
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with thoracic aorta dilatation | Baseline
  Thoracic aorta dilatation will be measured by TTE (Transthoracic echocardiogram). A value over 40 mm indicates thoracic aorta dilatation.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Newman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No